CLINICAL TRIAL: NCT01547429
Title: Artisan Aphakia Lens for the Correction of Aphakia in Adults
Brief Title: Artisan Aphakia Lens for the Correction of Aphakia (Secondary) in Adults
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Ophtec USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Artisan Adult Aphakia
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Aphakia
Keywords: aphakia; secondary intraocular lens
MeSH Terms: conditions — Aphakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraocular Lens Implantation for the Treatment for Aphakia (Experimental): Implantation of an Artisan intraocular lens to correct aphakia in Adults. No other information is needed to describe this section
  Interventions: Device: Artisan Aphakia Intraocular Lens

INTERVENTIONS:
Device: Artisan Aphakia Intraocular Lens — Implantation of lens to correct refractive error in aphakic eye

SUMMARY:
This study will determine the safety and effectiveness of the Artisan Aphakia Lens when used as a secondary implant to correct aphakia in adults.

DETAILED DESCRIPTION:
Not desired

ELIGIBILITY:
Inclusion Criteria:

* Patients 22 years of age and over at baseline visit of either sex and of any race where the natural lens has been removed or will be removed and a posterior chamber IOL is not indicated.
* Patient must agree to comply with the visit schedule and other requirements of the study

Exclusion Criteria:

* Patients that are not able to meet the extensive postoperative evaluation requirements
* Mentally retarded patients
* When the patient has no useful vision or vision potential in the fellow eye
* History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.), corneal dystrophy, degeneration, opacities or abnormalities that may affect vision.
* Abnormality of the iris or ocular structure which would preclude fixation, such as aniridia, hemiiridectomy, severe iris atrophy, rubeosis iridis, or other compromising iris pathology
* Patients with uncontrolled glaucoma
* High preoperative intraocular pressure, >25 mmHg
* Chronic or recurrent uveitis or history of the same
* Preexisting macular pathology that may complicate the ability to assess the benefit or lack of benefit obtained by the lens
* Patients with a retinal detachment or a family history of retinal detachment
* Retinal disease that may limit the visual potential of the eye such as retinopathy of prematurity or Stargardt's retinopathy Optic nerve disease that may limit the visual potential of the eye
* Diabetes mellitus
* Pregnant, lactating, or plans to become pregnant during the course of this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in best corrected visual acuity | 3 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Farhan, Study Director — Sponsor GmbH
Locations (18):
- United States (17):
  - Assil Eye Institute, Beverly Hills, California
  - Advanced Vision Care, Los Angeles, California
  - Yale Medicine Ophthalmology, Stratford, Connecticut
  - UF Health Eye Center, Gainesville, Florida
  - Price Vision Group, Indianapolis, Indiana
  - John Kenyon Eye Center, Jeffersonville, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Rosenthal Eye and Facial Plastic Surgery, Great Neck, New York
  - Pamel Vision and Laser Group, New York, New York
  - Sight MD, Rockville Centre, New York
  - New York Medical College, Westchester Medical Center, Valhalla, New York
  - Nevyas Eye Associates, Bala-Cynwyd, Pennsylvania
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - University of Tennessee, Hamilton Eye Clinic, Memphis, Tennessee
  - Focal Point Vision, San Antonio, Texas
  - Moran Eye Center, Salt Lake City, Utah
  - Valley Eye Associates, Appleton, Wisconsin
- Prism Eye Institute, Mississauga, Ontario, Canada